CLINICAL TRIAL: NCT00688285
Title: Automated Clinical Reminders in the Care of Chronic Kidney Disease Patients
Acronym: ACRinCKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Khaled Abdel-Kader, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PRO07110299
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; clinical alerts; late referral; electronic medical record; Computerized clinical decision support systems (CDSS)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): education and automated clinical alerts
  Interventions: Other: automated clinical alerts; Other: provider education
- 2 (Active Comparator): education session alone
  Interventions: Other: provider education

INTERVENTIONS:
Other: automated clinical alerts — automated clinical alerts in the electronic medical record
  Arms: 1
Other: provider education — PCP education session on CKD

SUMMARY:
To determine whether the use of educational sessions and computerized clinical reminders can improve primary care doctors' delivery of care to CKD patients compared to educational sessions alone. Hypothesis: Clinical reminders will improve the care delivered to CKD patients

DETAILED DESCRIPTION:
Literature supports that most chronic kidney disease (CKD) patients are cared for by primary care physicians (PCP) without the help of a kidney specialist. Many of these patients fail to achieve targeted outcomes and late referral to a nephrologist has been associated with an increased risk of death. Automated computerized clinical reminders have been shown to improve physician compliance with recommended guidelines in other settings.

Aims: To determine if clinical reminders can help PCPs decrease the rate of late referrals, improve urine albumin checks in CKD patients

Design: prospective randomized controlled, single-blinded study with additional historical control

Methods: Two 20-minute teaching sessions aimed at all GIM PCPs in the UPMC clinic followed by randomization of the eligible GIM providers to receive automated clinical reminders (CR) for their CKD stage 3b-5 patients versus routine care.

Outcomes: Using a database search, individuals with an eGFR<45ml/min/1.73m2 (not seen by a nephrologist) will have data collected on: PCP referral to a nephrologist, urinary albumin (or protein) quantification in the past year, PCP recognition of patients with eGFR<45ml/min, ACE/ARB usage.

ELIGIBILITY:
Inclusion Criteria:

* For PCPs: all GIM attending physicians with a weekly continuity clinic.
* For patients: >= 18 years-old with an eGFR<45ml/min/1.73m2 being seen in the UPMC GIM clinic by a faculty member during the 10-month intervention period

Exclusion Criteria:

* for PCPs: imminent plans to leave the department
* patients with a renal transplant, on any form of dialysis, or with a previous nephrology evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
referral to a nephrologist | 12 months
  Referral to a nephrologist within the 12 months following decision support system activation.

SECONDARY OUTCOMES:
Use of ACE/ARB | 12 months
  Active use of ACE/ARB at the end of the 12 month period following decision support system activation.
Annual ACR or PCR check | 12 months
  ACR or PCR within 12months of the decision support system activation

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Abdel-Kader, MD, Principal Investigator — University of Pittsburgh; Mark Unruh, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Abdel-Kader K, Fischer GS, Li J, Moore CG, Hess R, Unruh ML. Automated clinical reminders for primary care providers in the care of CKD: a small cluster-randomized controlled trial. Am J Kidney Dis. 2011 Dec;58(6):894-902. doi: 10.1053/j.ajkd.2011.08.028. Epub 2011 Oct 7. PMID 21982456